CLINICAL TRIAL: NCT04903691
Title: Changes in Fitness and Strength in Postoperative Cardiac Patients Undergoing Exercise Therapy: Biological and Functional Mechanisms of Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000028739
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Cardiorespiratory; Insufficiency, Due to A Procedure, Long-Term, Cardiac Surgery
Keywords: cardiorespiratory fitness

STUDY DESIGN:
Intervention Model Description: Intervention study with organized exercise program in intervention arm, no organized exercise in control arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): 130 patients who underwent open heart surgery and are cleared for exercise.These will include patients who enter supervised cardiac rehabilitation as well as patients who enter a supervised exercise program focusing strength training, endurance of functional training.
  Interventions: Behavioral: Cardiac Exercise Program
- Additional controls (No Intervention): 5 patients who choose not to enter any organized exercise program.

INTERVENTIONS:
Behavioral: Cardiac Exercise Program — Participants who enrolled in cardiac exercise program
  Arms: Exercise training

SUMMARY:
This study seeks to determine the biological, physiological and psychological effects of supervised exercise programs in patients surviving open heart surgery.

DETAILED DESCRIPTION:
Patients who have survived open heart surgery and cleared for exercise by their clinical team will be approached to enter a 12-week exercise program. Patient will consent to train with a personalized program either in strength, functional or aerobic exercise in a supervised setting for 3 sessions per week for a minimum of 12-week period. The aim is to enroll males and females in this arm in 1:1 ratio if possible. A separate cohort of patients entering cardiac rehabilitation (CR) will also be included for comparison. The CR program includes three sessions per week for a maximum of 36 sessions. The enrollment and retention rates in CR will be monitored. In this study, five patients who have undergone cardiac surgery and chosen not to participate in organized exercise program will be included. Participants cardiorespiratory fitness will be measured either using a questionnaire or in person. Through each phase of the study, the change in fitness, strength, biomarkers, body composition, cognition and psychosocial recovery will be monitored. All subjects will undergo detailed assessments in the research lab 2 weeks before and after finishing or exiting exercise program. A short (3-month) and long term (12-month) outcomes including rates of survival, major adverse cardiac events, cognition and cardiac-related hospitalizations will be collected as well during the study.

ELIGIBILITY:
Inclusion Criteria:

- Patients at least 18 years of age or older who undergo open heart surgery and who intend to enroll in a cardiac rehabilitation program.

Exclusion Criteria:

* Patients may be excluded for inability to read or understand English
* suffering from a condition that precludes informed consent (for example, cardiogenic shock)
* hemodynamic instability
* ongoing trauma or substance overdoses
* known intellectual or developmental delay
* communication impairment
* active users of illicit substances
* active psychiatric illness
* inability to attend cardiac rehabilitation (homeless, in police custody, or living out of state)
* inability to exercise (lower limb amputation, bedridden, decompensated heart failure, ongoing cancer treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness | Baseline and 2 weeks after completing exercise program
  Change in peak cardiorespiratory fitness as measured by metabolic equivalent (METS). (Higher values indicate higher fitness)
Change in strength | Baseline and 2 weeks after completing exercise program
  Change in strength as measured by grip strength (Higher values indicate better strength).
Change in functional fitness. | Baseline and 2 weeks after completing exercise program
  Change in functional fitness as measured by the Short Physical Performance Battery (higher overall score or less time to completion indicates higher fitness)
Change in cognition | Baseline and 2 weeks after completing exercise program
  Measured by standardized tests of cognition such as Montreal Cognitive Assessment (MoCA) (Higher values indicate better cognition with scores less than 23-26 adjusting for education indicative of impaired cognition)

CONTACTS AND LOCATIONS:
Overall Officials: Basmah Safdar, MD, Principal Investigator — Yale University
Locations (1):
- Yale Church Street Research Unit (CSRU), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided